CLINICAL TRIAL: NCT00441441
Title: A Randomized, Double-blind, Parallel Group Study Evaluating the Safety of Fluticasone Propionate/Salmeterol 100/50mcg HFA (2 Inhalations of 50/25mcg) Twice Daily Compared With Fluticasone Propionate 100mcg HFA (2 Inhalations of 50mcg) Twice Daily in Subjects 4-11 Years of Age With Persistent Asthma
Brief Title: A 12-Week Study To Assess The Safety Of Fluticasone Propionate/Salmeterol 100/50 Hydrofluoroalkane (HFA) Versus Fluticasone Propionate 100 HFA In Children With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFA106484
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: asthma; fluticasone propionate; children; fluticasone propionate/salmeterol
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone propionate/salmeterol 100/50 HFA (Experimental): Fluticasone propionate/salmeterol 100/50 HFA (2 inhalations of 50/25mcg), twice daily (strengths are ex-valve) and a placebo HFA inhaler matching the fluticasone propionate 100mcg HFA inhaler (2 inhalations) twice daily
  Interventions: Drug: fluticasone propionate/salmeterol
- Fluticasone propionate 100mcg HFA (Experimental): Fluticasone propionate 100mcg HFA (2 inhalations of 50mcg), twice daily (strengths are ex-valve) and a placebo HFA inhaler matching the fluticasone propionate/salmeterol 100/50 HFA inhaler (2 inhalations ) twice daily
  Interventions: Drug: fluticasone propionate

INTERVENTIONS:
Drug: fluticasone propionate — fluticasone propionate 100mcg HFA
  Arms: Fluticasone propionate 100mcg HFA
Drug: fluticasone propionate/salmeterol — fluticasone propionate/salmeterol 100/50mcg HFA
  Arms: Fluticasone propionate/salmeterol 100/50 HFA

SUMMARY:
This study is to assess the safety of an investigational drug in children 4 to 11 years of age who have asthma. The subjects will attend 7 clinic visits, of which up to 3 will be in the morning, and have lung function tests performed.

ELIGIBILITY:
Inclusion criteria:

* Must have asthma.
* Must be currently taking an inhaled corticosteroid.
* Must be able to attend 7 clinic visits, of which up to 3 will be in the morning, and have lung function tests that are at least 60% of normal (AM FEV1 or PEF).
* Have a historical or current FEV1 or PEF reversibility of >=12%.

Exclusion criteria:

* Has ever had life-threatening asthma (for example respiratory arrest, mechanical ventilation).
* Has a current ear or respiratory tract infection.
* Has ever had any other major illnesses (such as cystic fibrosis, heart problems, tuberculosis).

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 351 (Actual)
Dates: Start 2007-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (54):
- United States (19):
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Cortland, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, South Burlington, Vermont
- Australia (3):
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Subiaco, Western Australia
- Canada (4):
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Sarnia, Ontario
- Chile (3):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- GSK Investigational Site, San José, Costa Rica
- Germany (6):
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Gütersloh, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Wesel, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
- Latvia (2):
  - GSK Investigational Site, Ogre
  - GSK Investigational Site, Riga
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Utena
  - GSK Investigational Site, Vilnius
- Mexico (4):
  - GSK Investigational Site, Chihuahua City, Chihuahua
  - GSK Investigational Site, Monterrey N.L, Nuevo León
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- GSK Investigational Site, Lima, Lima Province, Peru
- Poland (2):
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Rabka-Zdrój
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Tomsk
- Spain (2):
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, San Javier (Murcia)

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Li JS, Qaqundah PY, Weinstein SF, LaForce CF, Ellsworth AV, Ortega HG, Ferro TJ. Fluticasone propionate/salmeterol combination in children with asthma: key cardiac and overall safety results. Clin Res Reg Affairs 2010;27(3):87-95.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: SFA106484 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SFA106484 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SFA106484 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SFA106484 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SFA106484 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SFA106484 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SFA106484 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 351 participants were enrolled in the study. However, only 350 of these 351 participants comprised the Intent-to-Treat Population, defined as all participants who were randomly assigned to treatment and received >=1 dose of Double-Blind study treatment.
Groups:
- Fluticasone Propionate/Salmeterol Hydrofluoroalkane (HFA): Participants who were randomly assigned to Fluticasone Propionate/salmeterol 100/50 micrograms (µg) HFA (2 inhalations of 50/25 µg), twice daily for 12 weeks.
- Fluticasone Propionate HFA: Participants who were randomly assigned to Fluticasone Propionate 100 µg HFA (2 inhalations of 50 µg), twice daily for 12 weeks.
Period: Overall Study
Arm/Group | Fluticasone Propionate/Salmeterol Hydrofluoroalkane (HFA) | Fluticasone Propionate HFA
Started | 173 | 177
Completed | 162 | 163
Not Completed | 11 | 14
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 4 | 6
Not completed — Exacerbation of asthma | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Fluticasone Propionate/Salmeterol HFA: Participants who were randomly assigned to Fluticasone Propionate/salmeterol 100/50 micrograms (µg) HFA (2 inhalations of 50/25 µg), twice daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA | Total
Number analyzed (Participants) | 173 | 177 | 350
Age, Customized [Number; unit: participants]
  4-5 years | 36 | 41 | 77
  6-11 years | 137 | 136 | 273
Gender [Count of Participants; unit: Participants]
  Female | 66 | 71 | 137
  Male | 107 | 106 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 73 | 143
  Not Hispanic or Latino | 103 | 104 | 207
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian/European Heritage | 114 | 113 | 227
  American Indian or Alaska Native | 24 | 27 | 51
  Central/South Asian Heritage | 8 | 8 | 16
  African American/African Heritage | 7 | 8 | 15
  Japanese Heritage | 3 | 0 | 3
  Arabic/North African Heritage | 2 | 2 | 4
  South East Asian Heritage | 2 | 0 | 2
  Mixed Race | 13 | 19 | 32

OUTCOME MEASURES:

1. Primary Outcome: Possible Drug-Related Adverse Events
Description: Adverse Events reported by the Investigator and judged by the Investigator to be possibly related to study drug, categorized by the Medical Dictionary for Regulatory Activities (MeDRA), were reported. ECG, electrocardiogram. QTc (corrected QT interval) and QT represent intervals on an ECG.
Time Frame: Treatment period (weeks 1-12) and Post Treatment (≥1 day after last time study drug)
Population: Intent-to-Treat (IITT) Population - All participants who were randomized and received at least one dose of double-blind study treatment.
Measure: Number; unit: participants
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
participants
  Participants with any drug-related event | 13 | 16
  Investigations - ECG QTc interval prolonged | 9 | 4
  Investigations - QT interval prolonged | 0 | 2
  Investigations - ECG QT borderline prolonged | 1 | 0
  Investigations - ECG QT interval abnormal | 1 | 0
  Cardiac - Defect conduction intraventricular | 2 | 7
  Cardiac - Conduction disorder | 1 | 1
  Cardiac - Sinus tachycardia | 1 | 0
  Cardiac - Supraventricular ectopics | 0 | 1
  Infections/Infestations - Oral candidiasis | 0 | 1
  Infections/Infest - Oropharyngeal candidiasis | 0 | 1
  Respiratory/thoracic/mediastinal - Dysphonia | 2 | 0

2. Primary Outcome: Investigator Evaluations of Electrocardiogram (ECG) Results
Description: ECGs were transmitted to an independent cardiologist who was responsible for providing interpretation of the ECG as either normal or abnormal (based on personal assessment). The investigator was then responsible for determining the clinical significance of the abnormal ECG in the context of the participants' history and clinical presentation. An abnormal, clinically significant ECG included, but was not limited to: prolonged QT interval, ischemic changes, ventricular hypertrophy, intraventricular conduction abnormalities, and clinically significant arrhythmias. PD, premature discontinuation.
Time Frame: Baseline and Week 12
Population: ITT Population. The number of participants at baseline was 173 and 177, respectively, for the Fluticasone propionate/salmeterol HFA and Fluticasone Propionate (FP) HFA groups. The number of participants at Week 12 was 162 and 160, respectively. Data for 6 participants in the FP treatment arm were either not obtained or not evaluable.
Measure: Number; unit: participants
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
participants
  Baseline - Normal | 145 | 155
  Baseline - Abnormal: Not Clinically Significant | 27 | 21
  Baseline - Abnormal: Clinically Significant | 1 | 0
  Week 12-No Change or insignificant Change | 136 | 142
  Week 12-Clinically Significant Change-Favorable | 2 | 0
  Week 12-Clinically Significant Change-Unfavorable | 24 | 18
  PD-No Change or insignificant Change | 7 | 9
  PD-Clinically Significant Change-Favorable | 0 | 1
  PD-Clinically Significant Change-Unfavorable | 0 | 1

3. Primary Outcome: Clinically Significant Unfavorable ECGs at Week 12
Description: Post-randomization ECGs categorized by the primary investigator as no change, significant change (favorable), significant change (unfavorable) from the ECG performed at Visit 1 (Baseline) are presented. Significant change (favorable) includes any ECG that improved from baseline, whereas significant change (unfavorable) includes any ECG that worsened from baseline. Clinical significance is determined by the primary investigator.
Time Frame: Baseline, Week 12
Population: ITT Population. The number of participants at baseline was 173 and 177, respectively, for the Fluticasone propionate/salmeterol HFA and Fluticasone Propionate (FP) HFA groups. The numbers of participants at Week 12 were 162 and 160, respectively. Data for 6 participants in the FP treatment arm were either not obtained or not evaluable.
Measure: Number; unit: participants
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
participants
  Clinically significant unfavorable change | 24 | 18
  AEs Reported for ECG findings | 22 | 18
  Clinically significant unfavorable ECGs repeated | 11 | 11
  Repeated ECGs w/ no change or insignificant change | 6 | 5

4. Primary Outcome: ECG Measures - Heart Rate
Description: The range of heart rates for this study was between 49-144 beats per minute
Time Frame: Baseline and Week 12
Population: ITT Population - All subjects who were randomized and received at least one dose of double-blind study treatment.
Measure: Mean (Full Range); unit: beats per minute
Groups:
- Fluticasone Propionate/Salmeterol HFA: Participants who were randomly assigned to Fluticasone propionate/salmeterol 100/50 micrograms (µg) HFA (2 inhalations of 50/25µg), twice daily for 12 weeks.
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
beats per minute
  Mean Heart Rate - Baseline | 84 [53 to 144] | 82.6 [51 to 136]
  Mean Heart Rate - Week 12 | 85.5 [59 to 138] | 81.9 [52 to 121]
  Mean Heart Rate - Premature Discontinuation | 73.1 [53 to 90] | 92.4 [49 to 130]

5. Primary Outcome: ECG Measures - QT Interval
Description: Fridericia's formula QTc interval=QT interval/cubed root of the R-R interval. The Bazett's formula QTc=QT/squared root of the R-R interval.
Time Frame: Baseline and Week 12
Population: ITT Population - All participants who were randomized and received at least one dose of double-blind study treatment.
Measure: Mean (Full Range); unit: milliseconds
Groups:
- Fluticasone Propionate HFA: Participants who were randomly assigned to Fluticasone propionate 100 µg HFA (2inhalations of 50 µg), twice daily for 12 weeks.
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
milliseconds
  Mean QTc Interval (Fridericia)- Baseline | 394.5 [340 to 449] | 390.8 [338 to 429]
  Mean QTc Interval (Fridericia) - Week 12 | 397.5 [355 to 439] | 393.6 [329 to 449]
  Premature Discontinuation (Fridericia) | 392 [359 to 417] | 394.8 [376 to 408]
  Mean QTc Interval (Bazett) - Baseline | 416.3 [356 to 464] | 411.4 [346 to 471]
  Mean QTc Interval (Bazett) - Week 12 | 420.8 [368 to 466] | 413.7 [351 to 477]
  Premature Discontinuation (Bazett) | 403.3 [376 to 446] | 422.7 [378 to 454]

6. Primary Outcome: Cardiovascular Adverse Events Reported During Treatment Period
Description: Cardiovascular Adverse Events, as categorized by the Medical Dictionary for Regulatory Activities (MeDRA), reported during Treatment Period. The Adverse Events were identified in any ECG interpretation by a central reader (Cardiologist) for any ECG obtained after the first treatment dose and were then reported by the Primary Investigator as an Adverse Event. Please see the category titles for a list of candidate cardiovascular adverse events.
Time Frame: 12-Week Treatment Period
Population: ITT Population - All participants who were randomized and received at least one dose of double-blind study treatment.
Measure: Number; unit: participants
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
participants
  Participants with Any Event | 98 | 103
  Electrocardiogram (ECG) Change | 3 | 2
  ECG QTc Interval Prolonged | 2 | 1
  ECG Abnormal | 1 | 1
  ECG QT Borderline Prolonged | 1 | 0
  Defect Conduction Intraventricular | 4 | 3
  Cardiac Arrhythmia | 1 | 0
  Premature Atrial Contraction | 1 | 0

7. Primary Outcome: Cardiovascular Adverse Events Reported During the Post-Treatment Period
Description: Cardiovascular Adverse Events, as categorized by the Medical Dictionary for Regulatory Activities (MeDRA), reported during Post-treatment period, defined as 1 day after last dose of study drug. The Adverse Events were identified in any ECG interpretation by a central reader (Cardiologist) for any ECG obtained after the first treatment dose and were then reported by the Primary Investigator as an Adverse Event.
Time Frame: 5 Days after Week 12
Population: ITT Population - All participants who were randomized and received at least one dose of double-blind study treatment.
Measure: Number; unit: participants
Groups:
- Fluticasone Propionate/Salmeterol HFA: Participants who were randomly assigned to Fluticasone Propionate/salmeterol 100/50 µg HFA (2 inhalations of 50/25 µg), twice daily for 12 weeks.
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
participants
  Participants with Any Event | 19 | 19
  ECG QTc interval prolonged | 11 | 5
  QT interval prolonged | 1 | 2
  ECG QT interval Abnormal | 1 | 0
  Defect Conduction Intraventricular | 2 | 7
  Conduction disorder | 1 | 1
  Sinus Tachycardia | 1 | 0
  Supraventricular Ectopics | 0 | 1

8. Primary Outcome: Asthma Exacerbations: Worsening of Asthma Requiring Emergency Intervention, Hospitalization, or Treatment With Asthma Medications Prohibited by the Protocols
Description: The Primary Investigator determined the severity of the exacerbation based on the participant's clinical presentation and the investigator's understanding of the disease, the participant, and his or her clinical experiences. The severity of the exacerbation was not defined in the protocol. Mild: Usually treated at home. Prompt relief with inhaled short-acting beta2 agonist. Possible short course of oral systemic corticosteroids. Moderate: Usually requires office or emergency department visit. Relief with frequent inhaled short-acting beta2 agonist. Oral systemic corticosteroids; some symptoms last for 1-2 days after treatment begins. Severe: Usually requires emergency department visit and likely hospitalization. Partial relief with frequent inhaled short-acting beta2 agonist. Oral systemic corticosteroids; some symptoms last for more than 3 days after treatment begins. Adjunctive therapies are helpful.
Time Frame: Treatment period (weeks 1-12)
Population: ITT Population - All participants who were randomized and received at least one dose of double-blind study treatment.
Measure: Number; unit: participants
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
participants
  Participants with any asthma exacerbation | 1 | 3
  Severity - Mild | 1 | 2
  Severity - Moderate/Severe | 0 | 1
  Withdrawal due to Asthma Exacerbation | 1 | 2

9. Primary Outcome: Number of Participants With the Indicated Levels of 24-hour Urinary Cortisol Excretion
Description: "Abnormal high cortisol excretion" and "Abnormal low cortisol excretion" are defined as above the upper limit of normal and below the lower limit of normal, respectively. The normal range for cortisol levels vary by age and gender. An abnormality is defined as a value of 24-hour urinary cortisol excretion that is outside the normal range. The normal range for 24-hour urinary cortisol excretion was provided by the central laboratory.
Time Frame: Baseline and week 12
Population: Cortisol Population - all participants not excluded due to the following reasons: missing data, use of protocol-specified corticosteroids (prior to screening), collection time outside of 24 ± 2 hours, use of inhaled cortical steroid (ICS) during treatment, and who stopped study medication >1 day prior to start of post-baseline urine collection.
Measure: Number; unit: participants
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 147 | 144
participants
  Baseline - Abnormal high cortisol excretion, n | 13 | 17
  Baseline - Abnormal low cortisol excretion, n | 1 | 0
  Week 12 - Abnormal high cortisol excretion, n | 13 | 8
  Week 12 - Abnormal low cortisol excretion, n | 2 | 0

10. Primary Outcome: Geometric Mean Values of 24-hour Urinary Cortisol Excretion at Baseline and Week 12
Description: Normal range for Cortisol levels vary by age and gender. Geometric mean is the product of the values taken to the Nth root, where N is the number of values in the set of values.
Time Frame: Baseline and Week 12
Population: Cortisol Population
Measure: Geometric Mean (Full Range); unit: Nanomoles per 24 hours (nmol/24 hrs)
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 147 | 144
Nanomoles per 24 hours (nmol/24 hrs)
  Baseline - Geometric Mean | 32.71 [2.7 to 156.2] | 30.88 [4.2 to 891.6]
  Week 12 - Geometric Mean | 25.03 [1.7 to 152.6] | 23.17 [5.3 to 145.8]

11. Primary Outcome: Geometric Mean Ratio for Week12:Baseline for 24-hour Urinary Cortisol Excretion
Description: Normal range for Cortisol levels vary by age and gender. The data provided are a direct calculation of the Week 12 geometric mean divided by the baseline value, nanomoles per 24 hours (nmol/24 hrs).
Time Frame: Baseline and Week 12
Population: Cortisol Population
Measure: Number; unit: ratio
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 147 | 144
ratio | 0.77 | 0.75

12. Primary Outcome: Number of Participants With the Indicated Levels of 24 Hour Urinary Cortisol Excretion by Spacer Use
Description: AeroChamber Plus spacers were provided for participants who demonstrated the inability to coordinate the use of an Meter Dose Inhaler at Visit 1. AeroChamber Plus spacer delivers 22% more medication than the original AeroChamber and is available in three mask sizes and without a mask. "Abnormal high cortisol excretion" and "Abnormal low cortisol excretion" are defined as above the upper limit of normal and below the lower limit of normal, respectively. An abnormality is defined as a value of 24-hour urinary cortisol excretion that is outside the normal range. The normal range for 24-hour urinary cortisol excretion was provided by the central laboratory.
Time Frame: Baseline and Week 12
Population: Cortisol Population
Measure: Number; unit: participants
Groups:
- Fluticasone Propionate/Salmeterol HFA - Spacer: Fluticasone propionate/salmeterol 100/50 micrograms (µg) HFA (2 inhalations of 50/25µg) twice daily in participants 4-11 years of age for 12 weeks - Participants who also used Spacers
- Fluticasone Propionate/Salmeterol HFA - No Spacer: Fluticasone propionate/salmeterol 100/50 µg HFA (2 inhalations of 50/25 µg) twice daily in participants 4-11 years of age for 12 weeks
- Fluticasone Propionate HFA - Spacer: Fluticasone Propionate 100 µg HFA (2 inhalation of 50 µg) twice daily in participants 4-11 years of age for 12 weeks. Participants who also used Spacers
- Fluticasone Propionate HFA - No Spacer: Fluticasone Propionate 100 µg HFA (2 inhalation of 50 µg) twice daily in participants 4-11 years of age for 12 weeks
Arm/Group | Fluticasone Propionate/Salmeterol HFA - Spacer | Fluticasone Propionate/Salmeterol HFA - No Spacer | Fluticasone Propionate HFA - Spacer | Fluticasone Propionate HFA - No Spacer
Number analyzed (Participants) | 115 | 32 | 113 | 31
participants
  Baseline - Abnormal high cortisol excretion | 12 | 1 | 14 | 3
  Baseline - Abnormal low cortisol excretion | 0 | 1 | 0 | 0
  Week 12 - Abnormal high cortisol excretion | 10 | 3 | 7 | 1
  Week 12 - Abnormal low cortisol excretion | 2 | 0 | 0 | 0

13. Primary Outcome: Geometric Mean Values of 24 Hour Urinary Cortisol Excretion by Spacer Use at Baseline and Week 12
Description: AeroChamber Plus spacers were provided for participants who demonstrated the inability to coordinate the use of an Meter Dose Inhaler at Visit 1. AeroChamber Plus spacer delivers 22% more medication than the original AeroChamber and is available in three mask sizes and without a mask. Geometric mean is the product of the values taken to the Nth root, where N is the number of values in the set of values.
Time Frame: Baseline and Week 12
Population: Cortisol Population
Measure: Geometric Mean (Full Range); unit: Nanomoles per 24 hours (nmol/24 hrs)
Groups:
- Fluticasone Propionate/Salmeterol HFA - Spacer: Fluticasone propionate/salmeterol 100/50 micrograms (µg) HFA (2 inhalations of 50/25 µg) twice daily in participants 4-11 years of age for 12 weeks - Participants who also used Spacers
Arm/Group | Fluticasone Propionate/Salmeterol HFA - Spacer | Fluticasone Propionate/Salmeterol HFA - No Spacer | Fluticasone Propionate HFA - Spacer | Fluticasone Propionate HFA - No Spacer
Number analyzed (Participants) | 115 | 32 | 113 | 31
Nanomoles per 24 hours (nmol/24 hrs)
  Baseline - Geometric Mean | 31.89 [3.6 to 156.2] | 35.84 [2.7 to 143.3] | 30.61 [4.2 to 891.6] | 31.89 [7.9 to 335.0]
  Week 12 - Geometric Mean | 23.37 [1.7 to 143.3] | 32.05 [4.6 to 152.6] | 23.20 [5.3 to 103.2] | 23.06 [5.4 to 145.8]

14. Primary Outcome: Geometric Mean Ratio for Week12: Baseline for 24 Hour Urinary Cortisol Excretion by Spacer Use
Description: AeroChamber Plus spacers were provided for participants who demonstrated the inability to coordinate the use of an Meter Dose Inhaler at Visit 1. AeroChamber Plus spacer delivers 22% more medication than the original AeroChamber and is available in three mask sizes and without a mask. The data provided are a direct calculation of the Week 12 geometric mean divided by the baseline value, nanomoles per 24 hours (nmol/24 hrs).
Time Frame: Baseline and Week 12
Population: Cortisol Population
Measure: Number; unit: ratio
Arm/Group | Fluticasone Propionate/Salmeterol HFA - Spacer | Fluticasone Propionate/Salmeterol HFA - No Spacer | Fluticasone Propionate HFA - Spacer | Fluticasone Propionate HFA - No Spacer
Number analyzed (Participants) | 115 | 32 | 113 | 31
ratio | 0.73 | 0.89 | 0.76 | 0.72

15. Secondary Outcome: Clinic Morning (AM) Forced Expiratory Volume in Participants 6-11 Years
Description: FEV1 (Forced Expiratory Volume in 1 second) is the volume of air that can be forced out in one second, after taking a deep breath. FEV1 is measured using a spirometer and obtaining "best effort" from 3 to 8 measurements. Week 12 is the measure taken at Week 12.
Time Frame: Baseline and week 12
Population: Subset of ITT Population: Participants who were 6-11 years of age (population not necessarily selected to show efficacy differences). Total numbers of participants analyzed for the Fluticasone propionate (FP)/salmeterol HFA and FP groups, respectively, were 137 and 136 at baseline; 126 and 124 at Week 12, and 6 and 7 at premature discontinuation.
Measure: Mean (Standard Error); unit: Liters per second (L/sec)
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 137 | 136
Liters per second (L/sec)
  Baseline - Mean FEV1 | 1.67 (0.035) | 1.64 (0.035)
  Week 12 - Mean FEV1 | 1.91 (0.038) | 1.82 (0.036)
  Week 12 - Mean Change from baseline | 0.24 (0.023) | 0.18 (0.023)
  Premature discontinuation - Mean FEV1 | 1.81 (0.14) | 1.70 (0.212)
  Premature discontin. - Mean Change from baseline | 0.03 (0.09) | -0.07 (0.120)

16. Secondary Outcome: AM Peak Expiratory Flow
Description: The peak expiratory flow (PEF) rate measures how fast a person can exhale air. It is used to compare to normal flow rates to predict obstruction and disease. The average PEF for a child or adolescent whose height is 43 inches is 147 Liters/minute (L/min), whose height is 66 inches is 454 L/min. Triplicate measurements taken for the best effort recorded.
Time Frame: Baseline and 12-Week Treatment Period
Population: Participants from the ITT Population (not necessarily selected to show efficacy differences). Total numbers of participants analyzed for the Fluticasone propionate (FP)/salmeterol HFA and FP groups, respectively, were 173 and 175 at baseline; 173 and 174 at Weeks 1-12; and 171 and 173 for the last 7 days on treatment.
Measure: Mean (Standard Error); unit: Liters/minute (L/min)
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
Liters/minute (L/min)
  Baseline - Mean AM PEF | 213 (4.83) | 203 (4.37)
  Weeks 1-12 - Mean AM PEF | 233 (5.07) | 220 (4.43)
  Weeks 1-12 - Mean Change from Baseline | 20.2 (2.04) | 17.4 (1.86)
  Last 7 Days on Treatment - Mean AM PEF | 238 (5.39) | 226 (4.73)
  Last 7 Days on Treatment-Mean Change from Baseline | 25.3 (2.58) | 23.3 (2.47)

17. Secondary Outcome: Asthma Symptom Scores
Description: Each morning prior dosing or PEF, self-scored based on past 24 hours: 0=No symptoms, 1=Symptoms for one short period, 2=Symptoms for two or more short periods, 3=Frequent Symptoms which did not affect activities of daily living (ADL), 4=Frequent.
Time Frame: Baseline and 12-Week Treatment Period
Population: Participants from the ITT population (not necessarily selected to show efficacy differences). Total numbers of participants analyzed for the Fluticasone propionate (FP)/salmeterol HFA and FP groups, respectively, were 173 and 175 at baseline; 172 and 174 at Weeks 1-12; and 167 and 170 for the last 7 days on treatment.
Measure: Mean (Standard Error); unit: Score in scale
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 177 | 173
Score in scale
  Baseline - Mean Score | 1.3 (0.06) | 1.4 (0.06)
  Weeks 1-12 - Mean Score | 0.9 (0.06) | 0.8 (0.05)
  Weeks 1-12 - Mean change from baseline | -0.4 (0.06) | -0.6 (0.06)
  Last 7 Days on Treatment - Mean Score | 0.8 (0.07) | 0.8 (0.07)
  Last 7 Days on Treat. - Mean change from baseline | -0.5 (0.07) | -0.6 (0.08)

18. Secondary Outcome: Percentage of Symptom Free Days
Description: Percentage of number of days without asthma symptoms based on Asthma Symptom Scores. Each morning prior to dosing or PEF, asthma symptoms were self-scored based on the past 24 hours: 0=no symptoms, 1=symptoms for one short period, 2=symptoms for two or more short periods, 3=frequent symptoms that did not affect activities of daily living (ADL), 4=frequent .
Time Frame: Baseline and 12-Week Treatment Period
Population: as for outcome 17
Measure: Mean (Standard Error); unit: Percentage of days
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
Percentage of days
  Baseline - Mean Percent | 20.0 (2.02) | 18.4 (2.00)
  Weeks 1-12 - Mean Percent | 46.7 (2.77) | 48.7 (2.80)
  Weeks 1-12 - Mean change from baseline | 26.8 (2.47) | 30.5 (2.62)
  Last 7 Days on Treatment - Mean Percent | 51.9 (3.51) | 53.4 (3.44)
  Last 7 Days on Treat. - Mean change from baseline | 32.1 (3.32) | 34.9 (3.43)

19. Secondary Outcome: Albuterol Use
Description: Albuterol inhalation aerosol was used as a rescue or prophylactic and recorded daily by subject or caregiver. The number of puffs of albuterol over the previous 24 hour period prior to dosing was recorded.
Time Frame: Baseline and 12-Week Treatment Period
Population: Participants from the ITT population (not necessarily selected to show efficacy differences). Total numbers of participants analyzed for the Fluticasone propionate (FP)/salmeterol HFA and FP groups, respectively, were 168 and 174 at baseline; 166 and 172 at Weeks 1-12; and 157 and 165 for the last 7 days on treatment.
Measure: Mean (Standard Error); unit: Number of puffs per 24 hours
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
Number of puffs per 24 hours
  Baseline - Mean number of puffs | 1.5 (0.12) | 1.8 (0.19)
  Weeks 1-12 - Mean number of puffs | 1.0 (0.09) | 0.9 (0.09)
  Weeks 1-12 - Mean change from baseline | -0.6 (0.12) | -1.0 (0.16)
  Last 7 Days on Treatment - Mean number of puffs | 0.7 (0.11) | 0.7 (0.11)
  Last 7 Days on Treat. - Mean change from baseline | 0.15 (0.8) | -1.2 (0.19)

20. Secondary Outcome: Percent of Albuterol-free Days
Description: Percentage of days when Albuterol use was unnecessary based on daily record and symptom free days.
Time Frame: Baseline and 12-Week Treatment Period
Population: as for outcome 19
Measure: Mean (Standard Error); unit: Percentage of days
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 173 | 177
Percentage of days
  Baseline - Mean percent rescue free | 43.7 (2.85) | 42.5 (3.04)
  Weeks 1-12 - Mean percent rescue free | 67.1 (2.46) | 70.0 (2.40)
  Weeks 1-12 - Mean change from baseline | 23.6 (2.79) | 28.3 (2.93)
  Last 7 Days on Treat. - Mean percent rescue free | 75.4 (2.96) | 75.8 (2.98)
  Last 7 Days on Treat. - Mean change from baseline | 30.4 (3.50) | 32.8 (3.58)

21. Post Hoc Outcome: Geometric Mean Values of 24-hour Urinary Cortisol Excretion at Baseline and Week 12
Description: A post-hoc analysis excluding participants with urine cortisol baseline values of >200 nanomoles/24 hours. Geometric mean is the product of the values taken to the Nth root, where N is the number of values in the set of values.
Time Frame: Baseline and Week 12
Population: Cortisol Population
Measure: Geometric Mean (Full Range); unit: Nanamoles per 24 hours (nmol/24 hrs)
Groups:
- Fluticasone Propionate/Salmeterol HFA: Samples provided by participants who were randomly assigned to Fluticasone Propionate/salmeterol 100/50 micrograms (µg) HFA (2 inhalations of 50/25 µg), twice daily for 12 weeks.
- Fluticasone Propionate HFA: Samples provided by participants who were randomly assigned to Fluticasone Propionate 100 µg HFA (2 inhalations of 50 µg), twice daily for 12 weeks.
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 147 | 140
Nanamoles per 24 hours (nmol/24 hrs)
  Baseline - Geometric Mean | 32.71 [2.7 to 156.2] | 28.39 [4.2 to 146.9]
  Week 12 - Geometric Mean | 25.03 [1.7 to 152.6] | 22.80 [5.3 to 145.8]

22. Post Hoc Outcome: Geometric Mean Ratio for Baseline:Week12 24-hour Urinary Cortisol Excretion
Description: A post-hoc analysis excluding participants with urine cortisol baseline values of >200 nmol/24 hrs. The data provided are a direct calculation of the Week 12 geometric mean divided by the baseline value, nanomoles per 24 hours (nmol/24 hrs) .
Time Frame: Baseline and Week 12
Population: Cortisol Population
Measure: Number; unit: ratio
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Number analyzed (Participants) | 147 | 140
ratio | 0.77 | 0.80

23. Post Hoc Outcome: Geometric Mean Values of 24-hour Urinary Cortisol Excretion by Spacer Use Excluding Participants With Abnormal Urinary Cortisol Excretion Values at Baseline From the Cortisol Population at Baseline and Week 12
Description: as for outcome 13
Time Frame: Baseline and Week 12
Population: Cortisol Population
Measure: Geometric Mean (Full Range); unit: Nanomoles per 24 hr (nmoles/24 hr)
Groups:
- No Spacer: Participants who did not use spacer and were in either treatment group
- Spacer: Participants who required a spacer and were in either treatment group
Arm/Group | No Spacer | Spacer
Number analyzed (Participants) | 58 | 202
Nanomoles per 24 hr (nmoles/24 hr)
  Baseline - Geometric Mean | 31.88 [7.9 to 81.7] | 27.08 [3.6 to 166.3]
  Week 12 - Geometric Mean | 27.85 [5.4 to 152.6] | 22.38 [1.7 to 143.3]

24. Post Hoc Outcome: Geometric Mean Ratio for Baseline: Week 12 24-hour Urinary Cortisol Excretion by Spacer Use Excluding Participants With Abnormal Urinary Cortisol Excretion Values at Baseline From the Cortisol Population
Description: AeroChamber Plus spacers were provided for participants who demonstrated the inability to coordinate the use of an Meter Dose Inhaler at Visit 1. AeroChamber Plus spacer delivers 22% more medication than the original AeroChamber and is available in three mask sizes and without a mask. The data provided are a direct calculation of the Week 12 geometric mean divided by the baseline value,nanomoles per 24 hours (nmol/24 hrs) .
Time Frame: Baseline and Week 12
Population: Cortisol Population
Measure: Number; unit: ratio
Groups:
- Spacer: Participants who did not use spacer and were in either treatment group
- No Spacer: Participants who required a spacer and were in either treatment group
Arm/Group | Spacer | No Spacer
Number analyzed (Participants) | 58 | 202
ratio | 0.87 | 0.83

ADVERSE EVENTS:
Arm/Group | Fluticasone Propionate/Salmeterol HFA | Fluticasone Propionate HFA
Serious Adverse Events (participants affected / at risk) | 1/173 | 0/177
Other Adverse Events (participants affected / at risk) | 61/173 | 68/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Propionate/Salmeterol HFA (N=173) | Fluticasone Propionate HFA (N=177)
Head Injury due to fall (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Propionate/Salmeterol HFA (N=173) | Fluticasone Propionate HFA (N=177)
Headache (Nervous system disorders) | 26 | 25
Upper Respiratory Tract Infection (Infections and infestations) | 11 | 13
Nasopharyngitis (Infections and infestations) | 16 | 21
Pharyngitis (Infections and infestations) | 4 | 12
Rhinitis (Infections and infestations) | 8 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Pyrexia (General disorders) | 8 | 16

LIMITATIONS AND CAVEATS:
A post-hoc evaluation confirmed that no clinically relevant ECG abnormalities were present. Differences in the primary and post-hoc analyses were associated with variation in the method of ECG interpretation and are not fully interpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.